CLINICAL TRIAL: NCT06585995
Title: Effectiveness and Safety of Two Vitamin D3 Supplementation Regimens in Adults with Early-stage COVID-19
Acronym: VDCOVID19ACUTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escuela Militar de Graduados de Sanidad, SEDENA (Other)
Responsible Party: Principal Investigator, IVÁN IGNACIO MEJÍA, Principal investigator, Escuela Militar de Graduados de Sanidad, SEDENA
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: No. 2022/C-015; No. 2022/C-015 (Other: EMGS)
Record Dates: First submitted 2024-08-21; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: COVID-19
Keywords: COVID-19; Cholecalciferol; Vitamin D; Interleukin-6; Glutathione peroxidase; Cough; dyspnea; fatigue; anxiety; depression
MeSH Terms: conditions — COVID-19; Cough; Dyspnea; Fatigue; Anxiety Disorders; Depression | interventions — Vitamin D; Cholecalciferol; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daily Vitamin D Supplementation Group (Experimental): This arm of the study involves daily administration of vitamin D to participants, with the dosage adjusted based on body weight and initial vitamin D levels, aiming to to investigate the efficacy of this regimen in improving vitamin D levels and reducing COVID-19 symptoms and IL-6, GPx and Von Willebrand Factor concentration.
  Interventions: Drug: vitamin D (cholecalciferol) supplementation
- Monthly Bolus Vitamin D Supplementation Group (Experimental): This arm of the study consists of administering a monthly bolus dose of vitamin D, equivalent to the total daily dose accumulated over the month, divided into 4 daily doses on 4 consecutive days, to investigate the efficacy of this regimen in improving vitamin D levels and reducing COVID-19 symptoms and IL-6, GPx and Von Willebrand Factor concentration.
  Interventions: Drug: vitamin D (cholecalciferol) supplementation

INTERVENTIONS:
Drug: vitamin D (cholecalciferol) supplementation — This pilot clinical study administered and compared daily and bolus vitamin D dosing regimens to achieve and maintain optimal serum 25(OH)D levels in patients with COVID-19. The daily dose group received constant cholecalciferol supplementation (vitamin D supplementation), aimed at achieving more stable and non-peak 25(OH)D levels. In contrast, the bolus group received a one-month cumulative monthly dose, divided into 4 doses, administered on 4 consecutive days, which could result in rapid increases followed by gradual decreases in 25(OH)D levels. The daily dose of cholecalciferol was calculated using the following formula: Daily dose of cholecalciferol = [Weight (kg) × desired increase in 25(OH)D (ng/ml) × 2.5] - 10 .
  Bolus dose = (daily dose)(30 days)/4 doses

SUMMARY:
This study aimed to determine the effectiveness and safety of individualized vitamin D3 supplementation in adult patients with early-stage severe COVID-19. The goal was to see if vitamin D3 could reduce the risk of progressing to critical COVID-19, characterized by severe respiratory distress and other life-threatening complications. The research question was: What is the effect of vitamin D3 on serum calcidiol levels during the active phase of the disease in adult patients with COVID-19?

The study hypothesized that an accelerated vitamin D3 supplementation regimen in adult patients with COVID-19 would achieve the ideal serum calcidiol level (40-60 ng/ml) during the active phase of the disease. This was a randomized controlled clinical trial with two parallel groups. The first group, the accelerated supplementation group, received a single monthly dose of vitamin D3, while the second group, the daily supplementation group, received a daily dose of vitamin D3 during their hospital stay. A total of 216 patients were included in the study and were randomly assigned to one of the two groups.

Key procedures and measurements included the collection of three blood samples from each patient during their hospital stay-at admission (day 1), on day 7, and on day 14. Biomarker analysis measured serum levels of vitamin D3, Von Willebrand Factor, interleukin-6 (IL-6), and glutathione peroxidase. Clinical monitoring was conducted to track the development of critical COVID-19, the need for mechanical ventilation, and overall clinical outcomes, such as recovery or death.

The importance of this study lay in the role of vitamin D3 in immune regulation, as it had been identified as a protective factor against severe respiratory infections. By determining the optimal supplementation strategy, this study hoped to improve clinical outcomes for COVID-19 patients, reduce mortality rates, and prevent the progression to critical illness.

Inclusion criteria for the study were adult patients aged 18-65 years with early-stage severe COVID-19, who had signed informed consent and had no contraindications for vitamin D3 supplementation. Exclusion criteria included patients with other severe comorbidities, those who were pregnant, those requiring immediate intensive care, and patients with a history of conditions that affect vitamin D metabolism.

Safety and efficacy monitoring tracked the vitamin D3 levels and correlated them with inflammation markers, oxidative stress, and thrombotic status to evaluate the impact of supplementation. Clinical progression was also monitored to assess the safety and efficacy of the vitamin D3 regimens.

Outcome measures included changes in serum calcidiol levels, correlation of calcidiol levels with biomarkers (IL-6, glutathione peroxidase, Von Willebrand Factor), duration and intensity of COVID-19 symptoms, incidence of critical COVID-19, need for mechanical ventilation, and overall clinical outcomes (recovery or death). This study aimed to provide valuable insights into the role of vitamin D3 in managing severe COVID-19, potentially informing treatment guidelines and improving patient outcomes.

DETAILED DESCRIPTION:
This randomized controlled clinical trial was designed to evaluate the effectiveness and safety of two vitamin D3 supplementation regimens in adult patients with early-stage severe COVID-19. The primary objective was to determine if vitamin D3 could help achieve optimal serum calcidiol levels (40-60 ng/ml) and reduce the risk of progressing to critical COVID-19.

The study included 216 adult patients who were diagnosed with early-stage severe COVID-19. Patients were randomly assigned to one of two groups. The first group, the accelerated supplementation group, received a single monthly dose of vitamin D3, while the second group, the daily supplementation group, received a daily dose of vitamin D3 during their hospital stay.

Each patient had three blood samples taken during their hospital stay to monitor the effects of vitamin D3 supplementation. The blood samples were collected at admission (day 1), on day 7, and on day 14. Each sample consisted of 7 ml of blood, with 2.5 ml used for serum analysis and 4.5 ml for plasma analysis. Biomarker measurements included serum levels of vitamin D3, Von Willebrand Factor, interleukin-6 (IL-6), and glutathione peroxidase. These biomarkers were measured using ELISA kits and analyzed via spectrophotometry. The vitamin D3 levels were quantified using the Vitros 5600 analyzer. The initial vitamin D3 measurement guided the calculation of the required dose for each patient.

Patients were closely monitored for the development of critical COVID-19, defined by severe respiratory distress requiring intensive care. Clinical monitoring included tracking the need for mechanical ventilation, defined by parameters such as PaO2 <60 mmHg, SpO2 <88%, and PaCO2 >50 mmHg with pH <7.32. The overall clinical outcomes, including recovery or death, were recorded. Any adverse events related to vitamin D3 supplementation were documented.

Clinical and laboratory data were collected systematically. Clinical data were gathered through collaboration with treating physicians and included detailed records of patient progression. Laboratory data were obtained from the hospital's pathology laboratory and stored securely. The blood samples were processed and stored in a biosecure environment, with serum and plasma components separated and stored in an ultracold freezer at -70°C until analysis.

Inclusion criteria for the study were adult patients aged 18-65 years with early-stage severe COVID-19, who had signed informed consent, and had no contraindications for vitamin D3 supplementation. Exclusion criteria included patients with severe comorbidities, such as terminal cancer or decompensated diabetes, pregnant or lactating women, patients requiring immediate intensive care, and patients with a history of conditions affecting vitamin D metabolism. Other exclusion criteria were recent use of high-dose vitamin D3 supplements, known intolerance to vitamin D3, and several other medical conditions that could interfere with the study.

Safety and efficacy were assessed by tracking serum vitamin D3 levels and correlating them with key biomarkers: inflammation (measured by IL-6 levels), oxidative stress (measured by glutathione peroxidase activity), and thrombotic status (measured by Von Willebrand Factor levels). Clinical outcomes and any adverse events were recorded throughout the study to determine whether vitamin D3 supplementation could positively influence these biomarkers and clinical outcomes.

The collected data were analyzed using a variety of statistical methods to ensure robustness. Descriptive statistics were used to summarize the data, including measures of central tendency (means, medians) and dispersion (standard deviations, ranges). The distribution of continuous variables was analyzed using Kolmogorov-Smirnov or Shapiro Wilks tests to assess the normality of the data. Pearson or Spearman correlation tests were used to evaluate the relationships between vitamin D3 levels and other biomarkers. Chi-square tests and T-tests or Mann-Whitney tests were used to compare proportions and means between the two groups. Survival analysis was performed using Kaplan-Meier curves and Cox proportional hazards models to assess the impact of biomarkers on patient survival. All statistical analyses were conducted with a significance level of p < 0.05, using PRISM v9.0 software.

Primary outcome measures included changes in serum calcidiol levels, correlations with biomarkers (IL-6, glutathione peroxidase, Von Willebrand Factor), and the duration and intensity of COVID-19 symptoms. Secondary outcome measures included the incidence of critical COVID-19, the need for mechanical ventilation, and overall clinical outcomes (recovery or death).

The study aimed to provide valuable insights into the role of vitamin D3 in managing severe COVID-19. By comparing two supplementation regimens, the study sought to identify the most effective strategy for achieving optimal vitamin D3 levels and improving patient outcomes. The findings could inform treatment guidelines and contribute to better clinical management of COVID-19, potentially reducing mortality rates and preventing the progression to critical illness.

ELIGIBILITY:
Inclusion Criteria:

1. Patients hospitalized for severe COVID-19 clinical presentation in the "early stage," with a maximum of 9 days after the onset of the first symptoms and who have not progressed to the "active phase" (fever, cough, sore throat, diarrhea, loss of taste or smell, oxygen saturation <92%, PaO2 / FiO2 <300 mmHg, respiratory rate >30 breaths per minute, or pulmonary infiltrates >50%).
2. Patients older than 18 years and younger than 65 years who have received at least 2 doses of the COVID-19 vaccine.
3. Patients who agree to participate at the time of hospitalization and sign the informed consent.
4. Patients with 25(OH)D levels below 40 ng/ml and without contraindications for Vitamin D3 supplementation.

Exclusion Criteria:

1. Patients who, at the time of recruitment, have another comorbidity as the primary condition for which they were hospitalized and that places them at high risk of death (e.g., terminal cancer, postoperative patients, renal failure, liver disease, uncontrolled diabetes, patients with HIV, CMV, tuberculosis, traumatic brain injury, shock from any cause, etc.).
2. Pregnant or breastfeeding patients.
3. Patients who have received Vitamin D3 supplements greater than 800 IU/day, 15 days before recruitment.
4. Patients with contraindications for Vitamin D3 supplementation, such as active granulomatous diseases (sarcoidosis, tuberculosis, lymphoma, Vitamin D3 metabolism disorders, hypercalcemia).
5. History of kidney stones.
6. Known Vitamin D3 hypervitaminosis or hypercalcemia.
7. Known intolerance to Vitamin D3.
8. Patients with extrapulmonary organ failure.
9. Patients with 25(OH)D levels equal to or greater than 40 ng/ml.
10. Patients who, at the time of recruitment, exhibit clear signs of "critical illness" due to COVID-19, such as organ failure requiring intensive care admission or who meet the criteria for mechanical ventilation due to oxygen desaturation: PaO2 <60 mmHg (after supplemental oxygen), SpO2 <88% (after supplemental oxygen), PaCO2 >50 mmHg with pH <7.32.

Elimination Criteria:

1. Patients who require major surgery after recruitment.
2. Patients who develop contraindications to standard COVID-19 treatment.
3. Patients who die before completing the three blood sample collections.
4. Patients who receive an IL-6 blocking drug.
5. Patients who develop clinical conditions that prevent blood sample collection or for whom medical recommendations advise against blood sample collection.
6. Patients who withdraw their consent to continue participating in the study.
7. Patients who develop adverse reactions secondary to Vitamin D3 administration, requiring the suspension of Vitamin D3, such as severe hypercalcemia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Glutathione Peroxidase (GPx) Activity | Baseline before supplementation, seven days and fourteen days after supplementation
  This measure evaluates the amount of glutathione peroxidase, such determination is performed by determining the glutathione peroxidase enzyme activity in the plasma of each patient, this parameter is determined with a special glutathione peroxidase enzyme activity determination kit, which indicates the bodys ability to reduce systemic oxidative stress. An increase in GPx activity is expected as a result of vitamin D supplementation.
Serum 25-Hydroxyvitamin D Levels | Baseline before supplementation, seven days and fourteen days after supplementation
  Vitamin D (calcidiol ) will be measured in each sample taken from each of the patients, this measurement will be performed by the clinical laboratory of the hospital center. This measurement will confirm the efficacy of the vitamin D supplementation regimen in achieving and maintaining sufficient serum vitamin D levels, the unit of measurement is nanograms/milliliters.
Serum Levels of Interleukin-6 (IL-6) | Baseline before supplementation, seven days and fourteen days after supplementation
  Interleukin-6 will be quantified in the serum of each patients sample using the ELISA technique. IL-6 is a proinflammatory cytokine. The study aims to observe changes in IL-6 levels, which could be significantly altered by vitamin D supplementation according to preliminary results.

SECONDARY OUTCOMES:
Intensity of headache | Baseline before supplementation, seven days and fourteen days after supplementation
  This measure will determine the intensity of the headache. And it will determine whether there is a significant association between vitamin D supplementation regimen and headache intensity.
Duration of fever in days | Baseline before supplementation, seven days and fourteen days after supplementation
  This measure will determine the duration (in days) of fever in each patient, this determination will be made by asking the patient if according to the body temperature in each day he/she presented or no longer presented a temperature higher than 38 degrees centigrade, the measurement will be made with a conventional thermometer. a sum of the days in which he/she did present fever (temperature higher than 38 degrees centigrade) will be made. Subsequently, this information will be used to determine whether there is a significant association between the vitamin D supplementation regimen and the duration of fever in days.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Pediatría, Mexico City, Mexico